CLINICAL TRIAL: NCT07321028
Title: Evaluation of In-Vitro Cryo Therapeutic Intervention on Human Cellular Samples - Truway Health Cryogenics Pilot Study
Brief Title: Evaluation of In-Vitro Cryo Therapeutic Protocols on Human Cell Samples (TWH-CRYO-001)
Acronym: CRYO-IVT
Status: Enrolling by invitation | Phase: Early Phase 1 | Type: Interventional
Sponsor: Truway Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TWH-CRYO-IVT-001
Record Dates: First submitted 2025-12-10; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Cellular Injury and Post-Cryogenic Recovery; Cryogenic Cellular Stress; Cold-Induced Cellular Injury; Thermal Injury Response; Post-Thaw Viability Impairment; Osmotic Stress Injury; Biomechanical Injury Modeling (In-Vitro); Blunt Force Injuries to the Extremities (Cellular Injury Model); Tissue Damage and Recovery Pathways; Hypothermic Tissue Stress; Cellular Regeneration and Repair
Keywords: Cryogenics; Cryopreservation; Freeze-Thaw Damage; Cellular Injury; Thermal Injury; Blunt Force Extremity Injury Model; In-Vitro Damage Response; Post-Thaw Regeneration; Osmotic Stress; Tissue Repair Pathways

STUDY DESIGN:
Intervention Model Description: Parallel assignment of human-derived cell samples into multiple intervention groups, including standard cryogenic freeze-thaw protocol, enhanced cryo-therapeutic protocol, and normothermic control. Each group is processed independently and concurrently to evaluate post-thaw viability, cellular injury response, and functional recovery.
Masking Description: This is an in-vitro laboratory protocol with no human participants. All interventions are openly assigned to specimen groups; therefore, no masking is required.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (3):
- Standard Cryopreservation Protocol (In Vitro) (Experimental): Human-derived cell samples are processed using a conventional laboratory cryopreservation protocol to establish baseline post-thaw viability and cellular recovery metrics.
  Interventions: Other: Standard Laboratory Cryopreservation Procedure
- Enhanced Cryotherapeutic Cryopreservation Protocol (In Vitro) (Experimental): Human-derived cell samples are processed using an optimized cryopreservation protocol designed to reduce cryo-induced cellular injury and improve post-thaw functional recovery.
  Interventions: Other: Enhanced Laboratory Cryopreservation Procedure
- Normothermic Cell Culture Control (No Cryopreservation) (Sham Comparator): Human-derived cell samples are maintained under standard normothermic cell culture conditions without exposure to freeze-thaw cycles to serve as a baseline control for cellular viability and function.
  Interventions: Other: Normothermic Cell Culture Control

INTERVENTIONS:
Other: Standard Laboratory Cryopreservation Procedure — Controlled-rate freezing of human-derived cell samples using an industry-standard cryoprotectant solution (10% dimethyl sulfoxide [DMSO] in culture medium) and defined cooling curves, followed by liquid nitrogen vapor storage and rapid rewarming. This intervention is conducted entirely in vitro for laboratory evaluation purposes only.
  Arms: Standard Cryopreservation Protocol (In Vitro)
Other: Enhanced Laboratory Cryopreservation Procedure — Modified in-vitro cryopreservation process incorporating alternative cryoprotectant formulations, optimized cooling rates, staged thawing procedures, and post-thaw recovery media adjustments. This protocol is investigational in nature but used solely for laboratory research and comparative performance assessment of cell preservation methods.
  Arms: Enhanced Cryotherapeutic Cryopreservation Protocol (In Vitro)
Other: Normothermic Cell Culture Control — Cells are cultured continuously under standard laboratory conditions without cryogenic exposure. No cryoprotectants, freezing, or thawing procedures are applied.
  Arms: Normothermic Cell Culture Control (No Cryopreservation)

SUMMARY:
This laboratory-based study evaluates the effects of controlled cryogenic preservation on human cell samples using Truway Health's in-vitro cryo therapeutic methodology. The study analyzes post-thaw viability, functional recovery, and morphological integrity following exposure to different cryopreservation parameters. Findings will support optimization of cryogenic protocols intended for future translational, biobanking, and therapeutic applications.

DETAILED DESCRIPTION:
Cryogenic preservation plays a central role in cellular therapy, long-term biological storage, regenerative medicine, and advanced manufacturing of therapeutic cell lines. This study investigates how varying cooling rates, cryoprotectant concentrations, and thaw-recovery procedures influence viability and functionality in human-derived cell samples.

The intervention consists of laboratory-controlled freeze-thaw cycles at temperatures ranging from -80 °C to -196 °C under defined standard and experimental conditions. Post-thaw evaluations include viability assays, growth kinetics, apoptotic markers, metabolic profiling, and structural assessment.

The study is non-clinical and does not involve living human subjects. All cell materials are obtained under appropriate consent or supplied as commercially available research-grade lines.

ELIGIBILITY:
Inclusion Criteria:

* This study does not enroll human participants. Eligibility applies only to human-derived cell samples.
* Samples must be de-identified prior to receipt.
* Samples must demonstrate ≥90% viability at pre-freeze assessment.
* Samples must be free of contamination (bacterial, fungal, mycoplasma).
* Samples must meet chain-of-custody and biospecimen compliance requirements.

Exclusion Criteria:

* No human participants will be enrolled or contacted.
* Any specimen containing identifiable private information.
* Samples with inadequate quality, contamination, or compromised viability.
* Samples obtained without appropriate donor consent or de-identification certification.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-12-10 (Actual); Primary Completion 2066-12-10 (Estimated); Study Completion 2066-12-10 (Estimated)

PRIMARY OUTCOMES:
Post-Thaw Viability | Twenty-four (24) hours after thaw
  Percentage of viable cells determined by trypan blue exclusion assay or automated cell viability analyzer.

SECONDARY OUTCOMES:
Cell Proliferation and Long-Term Viability at 7 Days | Seven (7) days after thaw
  Cell population doubling time and growth rate calculated from standardized growth curves generated under post-thaw culture conditions.
Apoptosis and Necrosis Marker Expression at 24 and 72 Hours | Twenty-four (24) hours and seventy-two (72) hours after thaw
  Percentage of cells positive for apoptosis or necrosis markers as determined by Annexin V / Propidium Iodide staining or caspase activity assays.
Cellular Metabolic and Functional Integrity from 24 Hours to 7 Days | From twenty-four (24) hours through seven (7) days after thaw
  Quantitative assessment of cellular metabolic activity and mitochondrial function using validated metabolic assays (e.g., MTT or resazurin reduction assays), and lineage-specific functional markers where applicable.
Morphological Integrity at 24 Hours | Twenty-four (24) hours after thaw
  Structural integrity and cellular morphology assessed by phase-contrast microscopy and scored using a predefined morphological grading scale.

CONTACTS AND LOCATIONS:
Overall Officials: Gavin Solomon, President & CEO, Principal Investigator — Truway Health, Inc.
Locations (1):
- Truway Health, Inc. , View 34, 401 E 34th Street, S11P, New York, NY 10016, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
This study does not involve human participants and does not generate individual participant data (IPD). All data are derived from in-vitro experiments using fully de-identified human-derived cell samples. Therefore, no IPD exists to be shared.

REFERENCES:
- See also: Truway Health, Inc. - Sponsor institution for CRYO-IVT protocol — https://www.truwayhealth.com
- See also: Introduction to cryopreservation principles and cellular responses to freezing — https://www.ncbi.nlm.nih.gov/books/NBK541103/